CLINICAL TRIAL: NCT06108908
Title: Influence of Inhaler Compliance on the Treatment of Asthma Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei Medical University Hospital (Other)
Collaborators: Taipei Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: N201905051
Record Dates: First submitted 2023-10-18; First posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Pulmonary Disease; Asthma
MeSH Terms: conditions — Lung Diseases; Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention Group: 1. Patients (compliance rate <80%) received active contact to remind on regular use of medication.
  2. The intervention is engaged in caring aspect behavior. None of regular asthma treatment is altered between groups.
  Interventions: Behavioral: Reminder
- Control: Patients were not informed regardless to their compliance rate.
  Interventions: Behavioral: Reminder

INTERVENTIONS:
Behavioral: Reminder — 1. The reminder is constrained in caring engagement that active engagements, e.g., phone call, or other instant messages, from study nurses to patients.

SUMMARY:
The major goal of "Influence of Inhaler Compliance on the Treatment of Asthma Patients" is to explore compliance rate outcome in adult asthmatic patients (20-80 years old) with mild to moderate persistent asthma according to American Thoracic Society (ATS) definition and diagnosis. The major endpoints include:

1. To increase the adherence rate of treatment by reminder intervention with correctly monitor patients' adherence rate by Asthma Supportive Kits
2. Eventually achieve best asthma care and management.

All participants will use Asthma Supportive Kits for 24 weeks and return visit on week 5, 12, 24. Based on collected data, the study compares intervention and control group to see if active reminder intervention may effectively alter compliance rate, and corresponding outcomes, e.g., asthma control status, acute exacerbation events.

DETAILED DESCRIPTION:
1. Upon enrollment, the all patients will be educated and equipped with asthma supportive kits, which is a electronic device attaches to an MDI medicine.
2. The asthma supportive kit registers every puff taken when the patient uses his/her MDI. The records are monitored by study nurses and calculated compliance ratio on rolling basis.
3. By enrollment, the patient is RANDOMLY assigned to Intervention and Control group. For the Intervention group in each study phases, when the given compliance ratio drops below 80% (as monitored by asthma supportive kit), the study nurse will actively engage to remind on medicine taking. For the Control group, the compliance ratio is calculated but to active engagement is applied.
4. All the patients adheres with regular asthma treatment mechanism, regardless to group assigned.

ELIGIBILITY:
Inclusion Criteria:

1. Adult asthmatic patients (20-80 years old)
2. With mild to moderate persistent asthma according to ATS definition and diagnosis
3. Willing to use Budesonide+Formoterol.
4. Adequately use inhaler
5. Without evident intentional non-adherence
6. Agree asthma is a common and potentially serious chronic disease
7. Willing to sign Informed Consent Form

Exclusion Criteria:

1. Inadequately use inhaler
2. Disagree asthma is a common and potentially serious chronic disease
3. With uncontrolled systemic diseases, such as hypertension, heart failure, renal failure, de-compensated liver cirrhosis, etc.;

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult asthmatic patients (20-80 years old) with mild to moderate persistent asthma according to ATS definition and diagnosis. Agree asthma is a common and potentially serious chronic disease.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-08-14 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
compliance ratio | 28 day
  Compliance Ratio:
  1. the Compliance Ratio evaluates the ratio of days which the patient is taking equal (or greater than) puffs of medicine as instructed by physician with the past 28-days.
  2. the outcome ratio ranges from 0% (none of days is taking correct amount) to 100% (all past 28 days were taking correct amount).
Asthma Control Test Score | 28 day
  Asthma Control Test (ACT) Score:
  1. the ACT is a patient self-administrated tool for identifying those with poorly controlled asthma;
  2. the test includes 5 items to recall past 4-week symptoms and daily functioning;
  3. The scores range from 5 as poorly controlled to 25 as completely controlled of asthma

CONTACTS AND LOCATIONS:
Overall Officials: Han-Pin KUO, Principal Investigator — Taipei Medical University, Taiwan, R.O.C.
Locations (1):
- Taipei Medical University, Taiwan, R.O.C., Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No